CLINICAL TRIAL: NCT03021941
Title: A MULTICENTER, OPEN LABEL, PHARMACOKINETICS, PHARMACODYNAMICS AND SAFETY STUDY OF ELELYSO(TM) (TALIGLUCERASE ALFA) IN PEDIATRIC SUBJECTS WITH TYPE 1 GAUCHER DISEASE
Brief Title: Pharmacokinetics, Pharmacodynamics And Safety Study Of Elelyso(tm) In Pediatric Subjects With Type 1 Gaucher Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: In a communication dated June 12, 2019 the FDA has released Pfizer from the Postmarketing Commitment (PMC 2767-2) that was associated with study B3031003.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B3031003
Record Dates: First submitted 2016-09-23; First posted 2017-01-16 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Gaucher Disease
Keywords: Gaucher Disease; Enzyme Replacement Therapy
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elelyso 60 units/kg (Other): All patients receive 60 units/kg of Elelyso.
  Interventions: Drug: Elelyso 60 units/kg

INTERVENTIONS:
Drug: Elelyso 60 units/kg — All patients receive Elelyso 60 units/kg.

SUMMARY:
In August of 2014, the FDA approved ELELYSO for long-term enzyme replacement therapy (ERT) for pediatric subjects with a confirmed diagnosis of Type 1 Gaucher disease. The recommended dosage for treatment-naïve adult and pediatric subjects 4 years of age and older is 60 units per kg of body weight administered every other week as a 60 to 120 minute intravenous infusion. As a postmarketing commitment, the Sponsor agreed to evaluate the pharmacokinetics (PK), pharmacodynamics (PD), and safety of Elelyso (taliglucerase alfa) in pediatric subjects with Type 1 Gaucher Disease. in at least 5 subjects with body weight less than 15 kg; at least 5 subjects with body weight 15 to less than 20 kg; and at least 5 subjects with body weight of 20-25 kg with Type 1 Gaucher disease dosed at 60 units/kg every other week.

When applicable, PD measurements for children enrolled in the PK study may be obtained through the taliglucerase alfa registry (PMR 1895-5) and will include organ volumes (spleen and liver), hematological values (hemoglobin and platelets) as well as growth (height and weight) data. Safety data, including any serious hypersensitivity reactions, such as anaphylaxis, as well as changes in antibody status (ie, detection and titers of binding and neutralizing antibodies, and detection of IgE antibodies), will also be collected through the taliglucerase alfa registry.

DETAILED DESCRIPTION:
This study (B3031003) is an open-label study in pediatric subjects with Type 1 Gaucher Disease to characterize PK, PD and safety following an infusion of taliglucerase alfa in at least 5 subjects with body weight less than 15 kg; at least 5 subjects with body weight 15 to less than 20 kg; and at least 5 subjects with body weight of 20-25 kg. The PK sample collection will take approximately 4 hours to complete and will be performed one month or up to 6 months after the subject's first taliglucerase infusion in the registry study. The subject will be contacted the day after the PK samples are collected to assess any continuing or new adverse events and to review the subject's concomitant medications. Body weight at the time of the PK blood draw will determine the weight category for each subject. Subjects enrolled into the study will be assigned the same unique subject number assigned to them in the registry study (B3031002). This will allow linkage to relevant data from the registry study for analysis in this study.

For the purposes of this study, baseline evaluations will be obtained from the registry study and must be performed prior to the subject's first dose of taliglucerase alfa. The Month 6 and Month 12 evaluations will be performed 6 months and 12 months after the start of taliglucerase alfa treatment, respectively.

Subjects will be eligible for the PK study (B3031003) only if the PD assessments (spleen volume/size, hemoglobin/platelet counts and height/weight measurements) immunogenicity data and Gaucher disease diagnostic history are available from the registry study baseline visit and prior to the start of taliglucerase alfa treatment. If liver volume/size is available, it will also be analyzed but is not necessary for eligibility for the PK study.

Pediatric subjects prescribed 60 units/kg of taliglucerase alfa every other week by their physician will be recruited from the registry study. Subjects can be screened for the PK study at the same time as they are enrolled into the registry study (ERT treatment-naïve subjects) or up to 6 months after they are enrolled into the registry study (previously ERT naïve subjects) if PD assessments (spleen volume/size, hemoglobin/platelet counts and height/weight measurements), immunogenicity data and Gaucher disease diagnostic history (residual enzyme activity and genotype data) were performed at baseline of the registry study and prior to the start of taliglucerase alfa treatment.

Baseline data from the registry study for PD and immunogenicity testing are defined as PD measurements (spleen volume/size, liver volume/size (if available), hemoglobin and platelet counts and growth measures), Gaucher disease diagnostic history and immunogenicity samples that were collected at entry into the registry study and prior to the start of taliglucerase alfa treatment.

For the secondary PD endpoints, spleen volume/size and liver volume/size (if available) will be measured using MRI, CT or ultrasound, whichever is the standard of care according to the investigator. The method used to measure spleen and liver volume/size at Baseline will be the same one used at Month 12. Change from Baseline and percent change from Baseline at Month 12 of registry study will be calculated for spleen volume, liver volume (if available), hemoglobin and platelet counts, and growth measures (height, weight and Z-scores).

For each subject enrolled in this study, safety data while on taliglucerase alfa, starting from the baseline visit (entry into the registry study) and continuing until 28 days after the Month 12 PD data collection visit, will be obtained for reporting.

Safety assessments for the study will include collection of all adverse event and serious adverse event data, including serious hypersensitivity reactions, procedures for immunogenicity testing (ie, detection and titers of binding and neutralizing antibodies and detection of IgE antibodies) as well as vital signs taken as standard of care during infusions. A pre-dose blood sample for testing of antidrug antibodies (ADA) on the day of PK Sample Visit will be collected in an effort to assess the impact of immunogenicity on PK.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric subjects with a diagnosis of Type 1 Gaucher disease (evidence of leukocyte acid-glucosidase activity 30% of the mean of the reference range for healthy persons), and meeting one of three weight categories: less than15 kg; 15 to less than 20 kg or 20-25 kg.
2. ERT treatment-naïve, or able to perform the PK assessment within the initial 6 months of initial Elelyso treatment (provided the subject was ERT naïve prior to the start of Elelyso).
3. Have had baseline (ie, prior to the first dose of study medication) PD measurements (spleen volume/size measured by MRI, CT or ultrasound, hemoglobin/platelet counts and growth measures including height and weight), immunogenicity sample collection and Gaucher disease diagnosis history documented in advance of treatment start.
4. Presence of splenomegaly at baseline defined as spleen volume/size measurement of 5 MN.
5. Subjects prescribed the nominal dose of 60 units/kg every two weeks and can tolerate an infusion rate of 1 mL/min.
6. Evidence of a personally signed and dated informed consent document from parent/legal guardian (or adult caregiver) capable of providing informed consent indicating that the subject's parent(s)/legal guardian has been informed of all pertinent aspects of the study before any screening procedures are performed. When age appropriate, written assent must also be obtained.
7. Have parent/legal guardian (or adult caregiver) capable and willing to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant issue or the presence of a medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator, would interfere with the subject's participation in the study, cause harm to the subject or decrease compliance with the study requirements.
2. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the PK sample collection visit, whichever is longer.
3. A diagnosis of Type 2 or 3 Gaucher disease, or the presence of neurological signs and symptoms characteristic of Type 2 or 3 Gaucher disease.
4. Any change during the registry study to the subjects dose of taliglucerase alfa infusion (ie, change from 60 units/kg every two weeks to a different dose of taliglucerase alfa) or a change in infusion duration or rate or a change of ERT medication (ie, switch from taliglucerase alfa to a different ERT).
5. In the judgment of the Investigator, the subject's vital signs (eg, blood pressure, pulse) prior to infusion on the day of the PK visit indicate that participation in the study would not be in the study candidate's best interest.
6. A hemoglobin level of <10 g/dL within 30 days of the PK sample visit or on the day of the PK sample visit.
7. History of sensitivity to heparin or heparin-induced thrombocytopenia. (Note: applies only if heparin lock or flush is to be used on the day of the PK sample visit).
8. Parents or legal guardians who are investigational site staff members directly involved in the conduct of the study and their family members, children of site staff members otherwise supervised by the Investigator, or subjects who are children of Pfizer employees directly involved in the conduct of the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - AUCinf | Up to 6 Months
  AUCinf of taliglucerase alfa assessed within 6 months from the subject's first dose of taliglucerase alfa.
Pharmacokinetics - AUClast | Up to 6 Months
  AUClast of taliglucerase alfa assessed within 6 months after the subject's first dose of taliglucerase alfa.
Pharmockinetics - Cmax | Up to 6 Months
  Cmax of taliglucerase alfa assessed within 6 months after the subject's first dose of taliglucerase alfa.
Pharmacokinetics - t½ | Up to 6 Months
  t½ of taliglucerase alfa assessed within 6 months after the subject's first dose of taliglucerase alfa.
Pharmacokinetics - CL | Up to 6 Months
  CL of taliglucerase alfa assessed within 6 months after the subject's first dose of taliglucerase alfa.
Pharmacokinetics - Vss | Up to 6 Months
  Vss of taliglucerase alfa assessed within 6 months after the subject's first dose of taliglucerase alfa.

SECONDARY OUTCOMES:
Pharmacodynamics - Spleen volume/size | 12 Months
  Spleen volume/size measured at Baseline and at Month 12.
Pharmacodynamics - Liver volume/size | 12 Months
  Liver volume/size measured at Baseline and at Month 12.
Pharmacodynamics - Growth measurements | 12 Months
  Growth measurements taken at Baseline and at Month 12.
Pharmacodynamics - Hemoglobin and Platelet Counts | 12 Months
  Hemoglobin and platelet counts measured at Baseline and at Month 12.
Safety - Antibody Assessment | 12 Months
  Antibody assessment measured at Month 6 and Month 12.
Safety - Adverse Events related to IV Infusion | 12 Months
  Adverse events related to intravenous infusions of taliglucerase alfa.
Safety - Vital Signs | 1 Day
  Vital signs prospectively collected during the taligluceras alfa infusion associated with PK measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- O&O Alpan LLC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3031003&StudyName=A+Multicenter%2C+Open+Label%2C+Pharmacokinetics%2C+Pharmacodynamics+And+Safety+Study+Of+Elelyso%28tm%29+%28taliglucerase+Alfa%29+In+Pediatric+Subjects+With+Type+1+Gaucher+Disease